CLINICAL TRIAL: NCT00005865
Title: A Research Study Evaluating Oral and Intravenous NAVELBINE as a Single Agent for the Treatment of Chemotherapy-Naive Subjects With Inoperable Stage IIIb or Stage IV Non-Small Cell Lung Cancer
Brief Title: Vinorelbine in Treating Patients With Stage IIIB or Stage IV Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000067897; GW-VINA2004
Record Dates: First submitted 2000-06-02; First posted 2004-03-24 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2007-06

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Vinorelbine

INTERVENTIONS:
Drug: vinorelbine tartrate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Giving drugs in different ways may kill more tumor cells. It is not yet known whether giving vinorelbine by mouth or infusion is more effective in treating non- small cell lung cancer.

PURPOSE: Randomized phase II trial to compare the effectiveness of vinorelbine given by mouth or as an infusion in treating patients who have stage IIIB or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the safety and efficacy of oral versus intravenous vinorelbine in patients with stage IIIB or IV non-small cell lung cancer. II. Compare the quality of life of patients treated with these regimens. III. Compare the pharmacokinetics of these treatment regimens in this patient population.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to one of two treatment arms. Arm I: Patients receive oral vinorelbine weekly. Arm II: Patients receive vinorelbine IV over 10 minutes weekly. Treatment continues in the absence of disease progression or unacceptable toxicity. Quality of life is assessed several times during treatment and 4 weeks after treatment. Patients are followed every 3 months for 1 year.

PROJECTED ACCRUAL: A maximum of 195 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed stage IIIB or IV non-small cell lung cancer not amenable to combination chemotherapy, curative surgery, or radiotherapy Bidimensionally measurable disease

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 60-100% Life expectancy: At least 12 weeks Hematopoietic: Granulocyte count at least 2,000/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 10 g/dL Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) SGOT less than 2.5 times ULN Alkaline phosphatase less than 5 times ULN (except in cases of bone or liver metastases) Renal: Creatinine no greater than 1.5 times ULN Cardiovascular: No unstable or uncontrolled cardiac disease Pulmonary: No history of recurrent aspiration pneumonitis within the past 3 months Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for 9 days after study Able to swallow capsules intact No active infection within the past 2 weeks No unstable or uncontrolled medical conditions No other prior malignancy within the past 5 years except basal cell skin cancer or carcinoma in situ of the cervix No history of peripheral neuropathy with severity greater than CALGB grade 1

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior immunologic therapy At least 1 week since prior hematopoietic growth factors or other blood products Chemotherapy: See Disease Characteristics No prior chemotherapy No other concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics At least 4 weeks since prior radiotherapy Surgery: See Disease Characteristics At least 2 weeks since prior surgery Other: At least 4 weeks since prior investigational device or drug No other concurrent anticancer therapy No other concurrent investigational device or drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-04; Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tess Delacruz, RN, BSN, Study Chair — GlaxoSmithKline
Locations (50):
- United States (46):
  - Arizona Clinical Research Center, Tucson, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Highlands Oncology Group, P.A., Fayetteville, Arkansas
  - Genesis Cancer Center, Hot Springs, Arkansas
  - NorthBay Healthcare System, Fairfield, California
  - Wilshire Oncology Medical Center, Pomona, California
  - Cancer Care Consultants of Northern California, Redding, California
  - Comprehensive Cancer Care Specialists of Boca Raton, Boca Raton, Florida
  - West Florida Cancer Institute - Pensacola, Pensacola, Florida
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - South Bend Clinic and SurgiCenter, South Bend, Indiana
  - Medical Oncology, LLC, Baton Rouge, Louisiana
  - Office of Luis Alberto Meza, Lafayette, Louisiana
  - Berkshire Physicians and Surgeons, P.C., Pittsfield, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - Lakeland Medical Center - St. Joseph, Saint Joseph, Michigan
  - Providence Hospital Cancer Center, Southfield, Michigan
  - St. Luke's Hospital, Duluth, Minnesota
  - Washington University Barnard Cancer Center, St Louis, Missouri
  - Mercy Oncology-Hematology Limited, St Louis, Missouri
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Trinitas Hospital - Jersey Street Campus, Elizabeth, New Jersey
  - Northern NJ Cancer Associates, Hackensack, New Jersey
  - Lovelace Health Systems, Albuquerque, New Mexico
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Office of Hal Gerstein, Great Neck, New York
  - Saint Vincents Comprehensive Breast Center, New York, New York
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - Veterans Affairs Medical Center - Northport, Northport, New York
  - University of Rochester Cancer Center, Rochester, New York
  - Office of Janak K. Choksi, Burlington, North Carolina
  - Raleigh Hematology/Oncology Associates - Wake Practice, Raleigh, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Ireland Cancer Center, Cleveland, Ohio
  - Hematology Oncology Consultants Inc, Columbus, Ohio
  - HillCrest Hospital, Mayfield Heights, Ohio
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - West Clinic, P.C., Memphis, Tennessee
  - Memphis Cancer Center, Memphis, Tennessee
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - Medical Group of Texas, Dallas, Texas
  - Joe Arrington Cancer Center, Lubbock, Texas
  - MultiCare Hematolgy/Oncology Clinic, Tacoma, Washington
- Canada (2):
  - Lakeridge Health Oshawa, Oshawa, Ontario
  - McGill University, Montreal, Quebec
- Puerto Rico (2):
  - Veterans Affairs Medical Center - San Juan, San Juan
  - University of Puerto Rico School of Medicine Medical Sciences Campus, San Juan

REFERENCES:
- [Result] Hirsh V, Desjardins P, Needles BM, Rigas JR, Jahanzeb M, Nguyen L, Zembryki D, Leopold LH. Oral versus intravenous administration of vinorelbine as a single agent for the first-line treatment of metastatic nonsmall cell lung carcinoma (NSCLC): A randomized phase II trial. Am J Clin Oncol. 2007 Jun;30(3):245-51. doi: 10.1097/01.coc.0000256103.21797.e5. PMID 17551300